CLINICAL TRIAL: NCT03867513
Title: MEGAbIT The Role of OPM MEG in Assessment and Diagnosis In mTBI. An Observational Study
Brief Title: The Role of MEG in Assessment and Diagnosis In mTBI
Acronym: MEGAbIT
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Other Study IDs: 19008; 256907 (Other: IRAS Project ID)
Record Dates: First submitted 2019-02-25; First posted 2019-03-08 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Brain Injuries, Traumatic
Keywords: Magnetoencephalography; Magnetic Resonance Imaging; Mild traumatic brain injury
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Concussion

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- mTBI cases: Those diagnosed with mild traumatic brain injury (mTBI) without abnormality on standard brain structural imaging, LOC ≤30mins, amnesia for ≤24hours, GCS ≥13 at all times and recovery to GCS 15 within 24hours)
  Interventions: Other: Multimodal imaging
- Acute trauma controls: Non-head trauma controls matched for age and sex with the mTBI group
  Interventions: Other: Multimodal imaging

INTERVENTIONS:
Other: Multimodal imaging — All participants will attend the Sir Peter Mansfield Imaging Centre for a scanning session using three imaging systems (SQUID MEG, OPM MEG and 7T MRI), cognitive testing and symptom questionnaires. Remote symptom monitoring and cognitive testing at three and six months.

SUMMARY:
Head injuries are responsible for 1.4 million visits to hospital each year in the United Kingdom (UK). Most patients are allowed home the same day and make a full recovery, but some will have persistent symptoms. The investigators aim to use the latest generation of imaging technology to investigate those with mild traumatic brain injury (mTBI) to better assess them.

The investigators will invite patients presenting following trauma to the Emergency Department at Queen's Medical Centre, Nottingham, UK to participate. The investigators will compare those who have a suffered an mTBI to those who have non-head traumatic injuries. The investigators will use two magnetoencephalogram (MEG) systems and ultra-high field magnetic resonance imaging (MRI) to record the functioning and structure of the brain within days of participants' injury. The investigators will test memory and thinking skills, then follow participants for six months, record the severity of participants' symptoms, and find out who does not make a full recovery.

Multimodal imaging will consist of a standard MEG device using Superconducting Quantum Interference Device (SQUID) sensors, a novel MEG device using Optically Pumped Magnetometer (OPM) sensors and seven Tesla MRI. The investigators will test whether these innovative imaging techniques are more sensitive to the acute damage that mTBI causes than routine imaging. The investigators will also test whether early imaging can reveal who is most seriously affected, identifying those who will not recover without additional support. It is currently not clear what the predominant mechanism of damage that causes these long-term problems is and the investigators hope this study will address this. The Medical Research Council is funding this work

ELIGIBILITY:
Inclusion criteria

* Participant is willing and able to give informed consent for participation in the study
* Male or female, aged 18-35
* In the Investigator's opinion, is able and willing to comply with all study requirements.
* Willing to allow his or her General Practitioner to be notified of participation in the study
* Two groups will be recruited:

  1. Diagnosed by the clinical ED team with mTBI (without abnormality on standard brain structural imaging, LOC ≤30mins, amnesia for ≤24hours, GCS ≥13 at all times and recovery to GCS 15 within 24hours)
  2. Diagnosed by the clinical ED team with non-head trauma, matched for age and sex with the mTBI group.

Exclusion criteria

* Patient requiring hospitalisation for ≥24 hours at presentation
* Any contraindication to undergo 7T MRI scan
* Pregnancy
* Other neurological, developmental or psychiatric disorders e.g. brain tumour, stroke, epilepsy, Alzheimer disease, schizophrenia, post-traumatic stress disorder, major depressive disorder, bipolar disorder or history of learning disability
* Previous hospital attendance with TBI
* Substance or alcohol abuse within six months of enrolment
* Taking certain medications thought to alter MEG signals: opioids and synthetic opioids (excluding codeine and dihydrocodeine), anti-epileptic drugs, sedatives, neuroleptics, and hypnotics
* Extensive metal dental hardware e.g. braces and large metal dentures (excluding fillings), implanted medical devices or other metal objects in the head, neck, or face areas that although they hold no risk to participants during a MEG recording may cause non-removable artefacts in the MEG data.
* Participants who have participated in another research study involving an investigational product in the past 12 weeks.
* Any other significant disease or disorder, which, in the opinion of the Investigator, may put the participants at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Potential participants will be identified form those attending the Emergency department of the Queen's Medical Centre, Nottingham
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-11-06 (Actual); Primary Completion 2021-05-05 (Estimated); Study Completion 2022-11-05 (Estimated)

PRIMARY OUTCOMES:
Can mTBI participants be differentiated from non-head injured controls by measuring brain wave activity? | Within two weeks of injury
  To measure and localize abnormal resting-state slow wave activity in an mTBI population in the acute stage (< 2 weeks post injury). Voxel-wise source reconstruction of MEG resting state data using a beamforming approach will be used to generate a normative database of brain activity in the cohort of age and sex matched non-head injured trauma participants. The investigators will compare the oscillatory power in the theta and alpha frequency band between the mTBI cohort and the normative database to generate statistical maps of abnormal brain activity on a per participant basis. These will be assessed for statistically significant loci of abnormal slow wave power.

SECONDARY OUTCOMES:
Is the SQUID or OPM MEG system preferred by participants for tolerability and ease of use? | Within two weeks of injury
  Participant preference for the SQUID or OPM MEG system will be recorded after both scanning sessions have been completed.

OTHER OUTCOMES:
What novel imaging measures best differentiate mTBI participants? | Assessment within two weeks of injury, follow up for six months
  To measure whole-brain connectivity in the resting state between regions defined via the automated anatomical labeling atlas. This will be achieved using amplitude envelope correlation between all signals originating from each region. Measures of node strength and overall connectivity will be calculated to investigate the efficiency of communication between brain regions in the participants' brains. The investigators will also measure structural connectivity using a diffusion tensor imaging (DTI) MRI sequence and structural damage using high-resolution susceptibility weighted imaging (SWI) MRI sequence. DTI will generate volumetric maps of fractional anisotropy.
Does abnormal slow wave activity on MEG arise from areas with SWI or DTI abnormalities? | Assessment within two weeks of injury, follow up for six months
  Compare per participant theta and alpha MEG power maps generated in the primary analysis with DTI and SWI MRI scans. Using volumetric quantitative techniques compare which MRI sequence better explains the variation in MEG signal.
Does early imaging provide prognostic information? | Assessment within two weeks of injury, follow up for six months
  Using a multivariate statistical model explore if baseline neuropsychological testing scores or memory task ability and symptom scales at six months correlate with baseline MEG and imaging abnormalities.
Is there a failure of the network responsible for attention switching in mTBI and is this correlated with objective deficits? | Assessment within two weeks of injury, follow up for six months
  Using a visual attention MEG protocol the investigators will assess participants' ability to switch their attention to different areas of their visual field during a task. The investigators anticipate the normally observed relative reduction in alpha and increase in gamma power over the contralateral occipital lobe will be disrupted in the mTBI participants compared to controls. The investigators hypothesis that this will be linked to worse task performance and they will compare whether both failure to modulate power and task performance are correlated with objective clinical measures.
Is there a failure of the network responsible for working memory in mTBI and is this correlated with objective deficits? | Assessment within two weeks of injury, follow up for six months
  Using an N-back working memory MEG protocol the investigators will assess participants' memory for worse task performance in the acute mTBI cohort and they will compare whether both MEG signal change and task performance are correlated with objective clinical measures.

CONTACTS AND LOCATIONS:
Overall Officials: Nikos Evangelou, MD, Principal Investigator — Clinical Neurology, Division of Clinical Neuroscience, University of Nottingham, UK
Locations (1):
- University of Nottingham, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided